CLINICAL TRIAL: NCT07154082
Title: A Prospective, Single-arm, Phase Ⅱ Study of Apatinib Mesylate and Camrelizumab Combined With TACE as Neoadjuvant Therapy for Resectable Centrally-located Hepatocellular Carcinoma in BCLC Stage B
Brief Title: Apatinib Mesylate and Camrelizumab Combined With TACE as Neoadjuvant Therapy for Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wei Zhang (Other)
Responsible Party: Sponsor-Investigator, Wei Zhang, Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-001
Record Dates: First submitted 2025-08-12; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: TACE; Hepatocellular carcinoma; Camrelizumab; apatinib; neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined with Camrelizumab and Apatinib (Experimental): Patients in the neoadjuvant treatment group will receive TACE treatment within one week after enrollment. One week after the resolution of the TACE treatment syndrome, they will be given Camrelizumab (200 mg, once every two weeks, for a total of 4 cycles) and oral Apatinib mesylate tablets (250 mg, once a day, for a total of 2 months).To ensure surgical safety, Camrelizumab should be discontinued at least two weeks before surgery, while Apatinib should be discontinued at least one week before surgery.
  Interventions: Drug: TACE (transarterial chemoembolization) combined with targeted/immunotherapy

INTERVENTIONS:
Drug: TACE (transarterial chemoembolization) combined with targeted/immunotherapy — Patients in the neoadjuvant treatment group will receive TACE treatment within one week after enrollment. One week after the resolution of the TACE treatment syndrome, they will be given Camrelizumab (200 mg, once every two weeks, for a total of 4 cycles) and oral Apatinib mesylate tablets (250 mg, once a day, for a total of 2 months).To ensure surgical safety, Camrelizumab should be discontinued at least two weeks before surgery, while Apatinib should be discontinued at least one week before surgery.

SUMMARY:
This study is a prospective, single-arm, phase Ⅱtrial. The subjects are patients resectable centrally-located hepatocellular carcinoma in BCLC stage B who are admitted to the Hepatobiliary Surgery Department of Tongji Hospital , Tongji Medical College, Huazhong University of Science and Technology, are over 18 years old, and have signed the informed consent form to voluntarily participate in this study. Through the neoadjuvant treatment of Apatinib mesylate and Camrelizumab combined with TACE before liver resection, it is expected to reduce the tumor size, lower the tumor burden, increase the surgical margin, improve the R0 resection rate, decrease the postoperative recurrence risk, and prolong the overall survival.

ELIGIBILITY:
Inclusion Criteria:

* 1) Diagnosed with hepatocellular carcinoma by pathological or histological examination.
* 2) the patient do not receive any anti-tumor treatment, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy and targeted therapy
* 3)resectable centrally-located hepatocellular carcinoma in BCLC stage B; Surgical resection was feasible after MDT discussion.
* 4) aged 18 to 70 years old, male or female
* 5) at least one measurable lesions (according to RECISTv1.1 requirements, The long diameter of the measurable lesion in the spiral CT scan is ≥10 mm or The short diameter of the enlarged lymph nodes is ≥15 mm)
* 6) ECOG score between 0 to 2, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤5 ULN, total serum bilirubin TBIL ≤1.5 ULN, creatinine (Cr)≤1.5ULN, HB≥80g/L, neutrophil > 1.5×109/L ,Serum albumin > 28 g/L
* 7) Child - Pugh grade A or B (7 points or less); ICG - R15 < 20%
* 8) Sufficient future liver reserve (FLR): For patients with liver cirrhosis, FLR should be greater than 40% of the standard liver volume; for patients without liver cirrhosis, FLR should be greater than 30% of the standard liver volume.
* 9) After assessment, TACE treatment can be deemed suitable.
* 10) The subjects signed the informed consent form and voluntarily received the neoadjuvant treatment of Apatinib mesylate and Carlimzumab combined with TACE. They had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* 1) Patients with intrahepatic cholangiocarcinoma (ICC), mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, or fibrolamellar hepatocellular carcinoma.
* 2) Patients with a history of malignant tumors other than liver cancer.
* 3) Patients with recurrent HCC after surgery who have received local or systemic treatment (chemotherapy, radiotherapy, surgery, interventional therapy, ablation, alcohol injection, or molecular targeted therapy).
* 4) Patients who are currently receiving or have previously received organ transplantation or allogeneic bone marrow transplantation, or have immune deficiency diseases or a history of organ transplantation.
* 5) Patients with vascular or biliary tumor thrombus or extrahepatic organ metastasis as shown by imaging.
* 6) Patients with moderate to severe ascites requiring therapeutic puncture and drainage or uncontrolled pleural effusion or pericardial effusion.
* 7) Patients with dysfunction of cardiovascular, respiratory, nervous, digestive, or urinary systems.
* 8) Patients with a history of gastrointestinal bleeding within 6 months before the start of the study, with a tendency to gastrointestinal bleeding, abdominal fistula, gastrointestinal perforation, or abdominal abscess.
* 9) Patients with multiple factors affecting oral drug administration (such as inability to swallow, chronic diarrhea, and intestinal obstruction, which significantly affect drug intake and absorption); patients allergic to the active ingredients or excipients of Camrelizumab and Apatinib mesylate.
* 10) Pregnant or lactating women; patients with reproductive capacity who are unwilling or unable to take effective contraceptive measures.
* 11) Patients with mental disorders or a history of abuse of psychotropic drugs.
* 12) Patients who have experienced thrombosis or embolism events within 6 months before the start of the study, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.
* 13) Patients without legal capacity or with restricted legal capacity.
* 14) Patients with any other conditions that the investigator deems unsuitable for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Two-year disease-free survival rate | From the time of undergoing the surgery to two years later
  DFS is defined as the time from surgical resection to local recurrence.

SECONDARY OUTCOMES:
ORR | The period from the onset of therapeutic effect until the confirmation of tumor progression，up to 24 months
  It refers to the proportion of patients whose tumors have shrunk to a certain extent and maintained that state for a certain period of time (mainly for solid tumors), including cases of complete response (CR, Complete Response) and partial response (PR, Partial Response).
MPR | max 24 months
  The residual surviving tumor tissue is ≤ 30%.
TTR | max 24 months
  TTR is defined as the time from the start of treatment until the first objectiveobservation of a response (either partia response, PR,or complete responseCR),provided that the response is subsequently confirmed
OS | max 24 months
  OS is defined as the time from study treatment to the date of death of thesubject, regardless of the cause of death.
DCR | max 24 months
  The proportion of patients who achieve complete response (CR) , partial response (PR) , or stable disease (SD) for a specified minimum duration according to standardized response criteria
R0 resection rate | max 24 months
  The proportion of cases where the tumor is completely removed and the microscopic margins are negative, meaning there is no tumor residue remaining.
AE | max 24 months
  Adverse events (AEs), Serious Adverse events (SAEs), surgery related safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China